CLINICAL TRIAL: NCT05449197
Title: Evaluation of the Evolution of the Patient Care Pathway in the Context of the Implementation of the DOuBLE EMIcizumab Dispensing Circuit in France
Brief Title: Evaluation of the Training Program for Community Pharmacists for Dispensing Emicizumab (HEMLIBRA®) in France
Acronym: PASODOBLEDEMI1
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1391
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Hemophilia A
Keywords: Haemophilia A; Accessibility; Emicizumab (HEMLIBRA®); Training evaluation
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community pharmacists chosen by the patient with haemophilia A for dispensing Emicizumab
  Interventions: Other: HEMOPHAR e-learning program

INTERVENTIONS:
Other: HEMOPHAR e-learning program — training on professional practice by following HEMOPHAR e-learning program

SUMMARY:
Haemophilia A (HA) is a rare constitutional haemorrhagic disease whose drug management is based on the use of chronic lifelong replacement therapy. The occurrence of an inhibitor is a dreaded complication that impacts conventional management, consisting in using factor VIII (FVIII)-based replacement therapy, most often for prophylaxis. Although effective, these treatments can only be administered intravenously, leading to accessibility constraints and significant mental burden for patients and their relatives.

Before June 15, 2021 in France, the emicizumab (HEMLIBRA®) was available only in hospital pharmacies for the prevention or reduction of bleedings. The introduction of the dual dispensing circuit in hospital or community pharmacies, left to patient's choice, is effective from this date. These changes have important organizational consequences for patients and health professionals alongside the pathway of care. Therefore, the effectiveness of this new organization requires to be evaluated with a national French study, called PASO DOBLE DEMI. The aims of this study are twofold :

I. To evaluate the direct impact of the training programs provided to the new placeholders of the dispensing circuit ; the community pharmacists, II. To evaluate satisfaction of patients or their relatives regarding the emicizumab treatment whether they chose dispensing in the community pharmacy, or kept the dispensing at the hospital pharmacy.

The methodology was based on the 4-level of the Kirkpatrick's evaluation model; 1) the immediate reaction of community pharmacists following the trainings (Reaction), 2) their knowledge acquisition (Learning), 3) their professional practice (Behavior) and 4 ) the patients' satisfaction related to their treatment whether dispensing in hospital or in community pharmacies (Results).

The PASO DOBLE DEMI I was based on the first three levels of the evaluation model.

ELIGIBILITY:
Inclusion Criteria:

* Pharmacists practicing in a pharmacy in metropolitan France
* Working in a pharmacy chosen by the patient with haemophilia type A
* And who have agreed to dispense Emicizumab (Hemlibra®)

Exclusion Criteria:

* Other pharmacy staff (including pharmacy technician, biologist, pharmacy students)
* Retired pharmacists at the date of the study
* Pharmacists who no longer practice in a community pharmacy dispensing Emicizumab (HEMLIBRA®)
* Pharmacists who expressed opposition to participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In March 2022, 300 community pharmacists have already followed-up the HEMOPHAR e-learning program, and the Laboratory Roche-Chugai counted approximately 450 community pharmacies which have ordered at least one time the treatment. We assumed that at least one pharmacist per community pharmacy followed the HEMOPHAR e-learning program, so with 2.5 pharmacists per community pharmacy, we estimated that 950 community pharmacists were concerned by dispensing Emicizumab (HEMLIBRA®) and potentially eligible for inclusion. This population was threefold depending on the training program followed-up (HEMOPHAR, Roche-Chugai) or absence of training program.
  With more than 2,500 hospital pharmacies throughout the metropolitan French territory, the hospital pharmacies met the pharmaceutical needs of people treated in health structures, medical and social structures. The eligible hospital pharmacists concerned all pharmacists practicing in hospital pharmacy on the date of the study.
Sampling Method: Non-Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Number of trained pharmacists dispensing emicizumab (HEMLIBRA (R)) in community pharmacies | 6 months.
Number of non-trained pharmacists dispensing emicizumab (HEMLIBRA (R)) in community pharmacies | 6 months.
Satisfaction of community pharmacists following the HEMOPHAR training program assessed by a likert scale | 6 months.
  levels of satisfaction (very satisfied,satisified, dissatisfied,very dissatisfied)
Professional practices of community pharmacists in dispensing emicizumab (HEMLIBRA (R)) assessed by a specific questionnaire | 6 months.
  specific questionnaire developed for the study

CONTACTS AND LOCATIONS:
Overall Officials: Valérie CHAMOUARD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chamouard V, Freyssenge J, Clairaz-Mahiou B, Ferrera Bibas F, Fraticelli L. Evaluation of an e-Learning Program for Community Pharmacists for Dispensing Emicizumab (Hemlibra) in France: Nationwide Cross-Sectional Study. JMIR Form Res. 2024 Apr 4;8:e54656. doi: 10.2196/54656. PMID 38574351
- [Derived] Fraticelli L, Freyssenge J, Prome-Combel E, Agnellet E, Dargaud Y, Chamouard V. Evaluation of the Care Pathway in the Context of the Dispensing of Emicizumab (Hemlibra) in Community Pharmacies in France: Protocol for a Cross-sectional Study Based on the Kirkpatrick Model. JMIR Res Protoc. 2023 Mar 8;12:e43091. doi: 10.2196/43091. PMID 36884286